CLINICAL TRIAL: NCT03026608
Title: Impact of a Public-Private Mobile Market to Improve Fruit & Vegetable Access
Brief Title: Green Cart Program Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: University at Buffalo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 12-1689
Record Dates: First submitted 2017-01-02; First posted 2017-01-20 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2016-12

CONDITIONS: Fruit and Vegetable Consumption; Food Insecurity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): Communities randomized to the intervention group receive the Veggie Van program shortly after randomization.
  Interventions: Behavioral: Veggie Van Program
- Delayed Intervention Control Group (Active Comparator): This group will receive the Veggie Van intervention approximately 6 months after baseline data collection and randomization (after the collection of 6 months outcomes data).
  Interventions: Behavioral: Veggie Van Program

INTERVENTIONS:
Behavioral: Veggie Van Program — This includes 1.) Weekly delivery of fresh local produce; 2.) Cooking and nutrition demonstrations; 3.) Weekly newsletters about cooking, nutrition and local produce mailed to all study participants and distributed at Veggie Van

SUMMARY:
The Green Car Evaluation was designed to test the impact of the Veggie Van mobile produce market on access to healthy food and fruit and vegetable intake in 12 lower-income communities using a cluster-randomized design.

DETAILED DESCRIPTION:
Lower-income and minority groups face significant health disparities with respect to obesity, cancer, heart disease and other chronic conditions. Poor diets, low in fruits and vegetables (F&V) and high in saturated fat, sodium and sugar, contribute to many of the health problems faced by vulnerable groups. While poverty, low-educational attainment and personal food preference are all associated with reduced F&V consumption, these individual-level factors must be viewed in an environmental context. Research has repeatedly demonstrated the important role that environment plays on health decisions and behaviors. Compared with higher-income neighborhoods, lower-income and minority neighborhoods are less likely to have a supermarket that sells a variety of F&V and other healthy foods. This is perpetuated by an underlying misconception that there is limited demand or potential profit for new healthy food ventures in these communities. In the few cases where new food outlets have opened in underserved areas, they have been met with substantial customer support. The NC Green Cart program, which our team has already been funded to lead, uses a weekly mobile market model to deliver low-cost boxes of fresh F&V to easily accessible community locations (such as churches and day care centers) and provide nutrition and cooking education. This program builds upon burgeoning support for a local sustainable food system in NC and leverages a public-private partnership to increase access to fresh F&V in underserved communities. While current program funding allows for minimal evaluation, the present study hopes to demonstrate that selling affordable, accessible F&V in lower-income communities is not only financially viable, but can impact behavioral risk factors of individuals in target communities. Working together with the Green Cart program team, this research will 1.) measure the impact of a mobile market at 6, 12 and 18 months on the primary outcome of F&V consumption as well as BMI, perceived access to F&V, and self-efficacy to purchase, prepare, serve and eat fresh F&V using a randomized controlled design; and 2.) assess community support, feasibility, and financial sustainability of the public-private Green Cart partnership. Results of this research will inform our understanding of how the food environment impacts dietary choices and provide evidence for researchers, businesses, non-profits and policy makers on the potential impact and viability of using similar models to reduce food access disparities and improve diet.

ELIGIBILITY:
Inclusion Criteria:

* Receives services or lives within one of the communities selected for the study
* Main shopper for the household
* Intends to use Veggie Van if it comes to their community

Exclusion Criteria:

* Under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2012-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change in Fruit and Vegetable Consumption | Change from baseline to 6 months
  Measured via food frequency questionnaire

SECONDARY OUTCOMES:
Change Score for Perceived access to fresh fruits and vegetables | Change from baseline to 6 months
  At each time point, a three-question perceived access scale was used to measure participants' perceptions of access to fresh fruits and vegetables in (1) their neighborhood, (2) the area surrounding the VV community site, and (3) in general. Questions included 1) "It is easy to buy fresh fruits and vegetables [in my neighborhood/around community sites/ in general];" 2) "There is a large selection of fresh fruits and vegetables [in my neighborhood/around community site/in general];" 3) "The fresh fruits and vegetables [in my neighborhood/around community site/in general] are high quality." For all perceived access questions, participants chose responses from a 5-point Likert scale ranging from "Strongly Agree" = 5 to "Strongly Disagree" = 1. Each three item scaled was summed to create a perceived access score by location (range 3-15). Higher scores at each time point indicate higher perceived access and positive changes indicate increases in access from baseline to 6 months.

OTHER OUTCOMES:
Change in Body Mass Index | Change from baseline to 6 months
  measured via self-reported height and weight

CONTACTS AND LOCATIONS:
Overall Officials: Alice Ammerman, PhD, Principal Investigator — University of North Carolina, Chapel Hill

IPD SHARING:
Plan to Share IPD: No
No plan to share individual data

REFERENCES:
- [Derived] Leone LA, Tripicchio GL, Haynes-Maslow L, McGuirt J, Grady Smith JS, Armstrong-Brown J, Gizlice Z, Ammerman A. Cluster randomized controlled trial of a mobile market intervention to increase fruit and vegetable intake among adults in lower-income communities in North Carolina. Int J Behav Nutr Phys Act. 2018 Jan 5;15(1):2. doi: 10.1186/s12966-017-0637-1. PMID 29304862